CLINICAL TRIAL: NCT00474565
Title: Contrast-Enhanced Coronary Artery and Coronary Artery Bypass Graft Imaging Using Aortic Root Catheter Injection With Computed Tomographic Angiography (CTA)
Brief Title: Coronary Artery and Coronary Artery Bypass Graft Imaging Using a Specialized Catheter and Computed Tomography
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended failure to follow Conflict of Interest Management Plan
Sponsor: Corewell Health East (Other)
Responsible Party: Nishit Choksi, M.D./Principal Investigator/Interventional Cardiologist, William Beaumont Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2005-156
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease
Keywords: Catheter,; Aortic root injection,; low dose contrast injection,; coronary artery angiogarm and; coronary artery bypass graft imaging.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Placement of an aortic root pigtail catheter. — Seldinger technique for placement of catheter.

SUMMARY:
The present study relates to a new approach to coronary artery and coronary artery by-pass graft imaging, and more particularly to computed tomographic angiography following an aortic root injection of a low amount of contrast (up to 30 cc) via a percutaneously placed catheter (Vanguard DX, Medrad Inc.) positioned in the aortic root.

The objective of the study is to show the feasibility of Coronary artery CTA using aortic root injection of contrast compared to the standard invasive cardiac catheterization.

DETAILED DESCRIPTION:
Coronary artery disease remains the leading cause of death worldwide. The diagnosis via the gold standard, cardiac catheterization, remains a time consuming, expensive, and invasive procedure with some considerable risks. In addition, there is a significant risk due to cumulative amount of iodinated contrast delivered (between 80 - 120 cc) in patients who have abnormal renal insufficiency or at a high risk for developing contrast nephropathy. Cardiac catheterization specifically involves arterial puncture with a needle, usually in the groin or upper extremity, through which a guidewire is passed fluoroscopically to the ascending aorta. A catheter is then inserted over the guidewire and subsequently, the guidewire is removed and iodinated contrast is injected to opacify the aorta or coronary arteries. As such, there are different kinds of catheters that are used to engage either the right or left native coronary arteries or by-pass vein grafts. This procedure requires separate injections into the coronary arteries or by-pass grafts which can induce arrhythmias, require over one hour of procedural time, requires larger bore catheters, exposes the physician and patient to ionizing radiation and subjects the patient with coronary artery disease to contrast induced nephropathy, especially in cases requiring higher loads of iodinated contrast.

Of the noninvasive techniques, the most common limiting factor when employing IV-enhanced CTA is the underlying blood pool, which also enhances when contrast-enhanced protocols are employed using a peripheral intravenous contrast injection route. This results in a frequent obscuration of the native coronary arteries. Reproducible enhancement of the distal and tributary anatomy is another pitfall with IV-enhanced coronary CTA. In addition, the amount of contrast agent required is similar to that amount required during invasive coronary angiography. As such, the method of the present study provides an imaging concept of the coronary arteries employing a catheter device in conjunction with computed tomography (CT) imaging machine that will enable a reduction of the total amount of dye delivered to the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients that have an abnormal nuclear medicine heart scan and are already scheduled for cardiac catheterization for evaluation of coronary artery disease or disease of coronary artery bypass grafts will be asked to participate in this trial.
2. Provided informed consent.
3. Evaluation by a Cardiology Division staff or Cardiology nurse clinician.

Exclusion Criteria:

1. Patient is currently enrolled in another related research study.
2. Less than 18 years of age.
3. Pregnant patients.
4. Abnormal renal function with creatinine equal to or greater than 1.6 mg/dl or those subjects requiring dialysis.
5. Patients with chronic obstructive pulmonary disease or heart-failure with cardiac ejection-fraction less than 30%.
6. Patients with known sensitivity to beta-blockers (Lopressor) or have asthma.
7. Patients receiving an abnormally large volume of contrast media during cardiac catheterization (> 200cc)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Coronary artery diameters and degree of stenosis are assessed and compared between conventional cath angio and new CTA study. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abbas, M.D., Study Director — Corewell Health East; Kostaki G. Bis, M.D., Study Chair — Corewell Health East; Nishit Choksi, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, 3601 West 13 Mile Road, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Kumar A, Bis KG, Shetty A, Vyas A, Anderson A, Balasubramaniam M, O'Neill W, Stein W. Aortic root catheter-directed coronary CT angiography in swine: coronary enhancement with minimum volume of iodinated contrast material. AJR Am J Roentgenol. 2007 May;188(5):W415-22. doi: 10.2214/AJR.06.0945. PMID 17449736